CLINICAL TRIAL: NCT05598099
Title: Concentrated Exposure Therapy for Post-traumatic Stress Disorder - a Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: B4DT-PTSD1
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: PTSD
Keywords: CBT; CAPS; Group therapy; Psychotherapy; Treatment satisfaction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individual therapy over four consecutive days: Treatment will be delivered individually over four consecutive days
  Interventions: Behavioral: Concentrated cognitive behavioral therapy
- Combined Individual and group therapy over four consecutive days: Treatment will be delivered in a mix of individual and group sessions over four consecutive days
  Interventions: Behavioral: Concentrated cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Concentrated cognitive behavioral therapy — A psychological intervention consisting of psychoeducation and exposure therapy with the goal of changing the tolerability and negative interpretations of post-traumatic symptoms. The treatment is tailored to the individual patient through all stages, including relapse prevention and planning how to use treatment principles in daily life
  Other Names: Bergen 4-Day Treatment

SUMMARY:
Post-traumatic stress disorder (PTSD) is a prevalent and disabling condition. Trauma-focused psychotherapy, including cognitive behavioural therapy (CBT), are among the recommended first-line treatment alternatives. However, a substantial proportion of patients decline, drop-out or do not respond to current psychotherapies. Previous research suggests that intensive or concentrated formats of trauma-focused psychotherapy can lead to faster recover and lower attrition, but there are currently few studies of these approaches. The current study will investigate the acceptability. treatment satisfaction and preliminary changes in symptoms after four consecutive days of concentrated CBT for PTSD.

DETAILED DESCRIPTION:
The study will investigate the research questions in three stages. In the first stage four patients will be treated individually. In the second stage two groups of four patients will be treated, with at least a 1:1 ratio between therapists and patients per group. In the third stage 30 patients will be treated in groups of about four patients per group, with at least a 1:1 ratio between therapists and patients per group. The primary outcome measure is changes in PTSD-related symptoms as measured using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Acceptability will be measured as the proportion of patients accepting treatment when offered, while attrition is measured as the proportion of patients that withdraw from treatment after it has started. Several other measures will be collected to measure treatment satisfaction, related symptoms, and functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* fulfills DSM-5 criteria for PTSD
* One or more single traumas in adolescence or adulthood
* Speaks and writes Norwegian

Exclusion Criteria:

* New or unstable psychopharmacological treatment within last four weeks
* fulfills ICD-11 criteria for complex PTSD
* Ongoing substance abuse
* Ongoing danger of suicide
* Ongoing borderline personality disorder
* Ongoing psychosis
* Intellectual disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with PTSD recruited from clinics and popular media referred to Clinic for 4-Day Treatment at Haukeland University Hospital, Bergen, Norway
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change in scores from before treatment to one week after treatment
  Clinician-administered interview to diagnose and the severity of PTSD
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change in scores from one week after treatment to three months after treatment
  Clinician-administered interview to diagnose and the severity of PTSD
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change in scores from three months after treatment to twelve months after treatment
  Clinician-administered interview to diagnose and the severity of PTSD

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire 8 (CSQ-8) | One week after treatment
  Patient-rated questionnaire of treatment satisfaction
Client Satisfaction Questionnaire 8 (CSQ-8) | Three months after treatment
  Patient-rated questionnaire of treatment satisfaction
Client Satisfaction Questionnaire 8 (CSQ-8) | Twelve months after treatment
  Patient-rated questionnaire of treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Anders L Thorsen, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not planned